CLINICAL TRIAL: NCT04474886
Title: Intervention With Oral Nutritional Supplement (ONS) for the Patient With or at Risk of Malnutrition
Brief Title: Oral Nutritional Supplement for the Patient With or at Risk of Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Timothy Kwok, professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020.223
Record Dates: First submitted 2020-07-09; First posted 2020-07-17 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresubin® powder fibre (Experimental): 2 servings of Fresubin® powder fibre per day as supplement to normal diet
  Interventions: Dietary Supplement: Fresubin® powder fibre
- Usual diet (No Intervention): Maintain usual diet

INTERVENTIONS:
Dietary Supplement: Fresubin® powder fibre — 2 servings per day
  Arms: Fresubin® powder fibre

SUMMARY:
In case of acute and chronic illness nutritional problems are widespread, and a reduced dietary intake in combination with effects of catabolic disease rapidly lead to malnutrition. A high prevalence of protein energy malnutrition in patients has been reported. A close relation between malnutrition and re-admission rate, cost of hospital care in terms of length of stay in hospital as well as mortality has been documented. A Cochrane review of the use of oral nutritional supplementation suggested that oral nutrition not only provided nutrients, but also has significant improvements on psychological and social functions, possibly through enhancing sensation of taste and flavor which is an important mediator of pleasure and well-being. Therefore, an oral option of nutrition is always considered as the first choice of nutritional intervention, in particular in situations where nutritional interventions, such as assisted feeding, are difficult, time-consuming and demanding due to advanced morbidity and slow responses. In this randomized controlled trial, the investigators will explore the gaps of nutritional needs and the potential use of nutrition supplementation in the management of malnutrition among patients in Hong Kong. The investigators aim to improve the nutrient intakes and the nutritional status of participants through a specially formulated oral nutrition supplement titled "Fresubin® Powder Fibre" to reverse malnutrition status due to acute and chronic illness. Fresubin® Powder Fibre is a nutritionally complete powder product to be reconstituted in different caloric densities (1.0 to 1.5 kcal/ml) and containing high quality protein and vitamin D for the dietary management of participants with or at the risk of malnutrition.

ELIGIBILITY:
Inclusion Criteria:

* Chinese origin aged 18 or above
* Normally reside in Hong Kong
* Could speak and understand Chinese
* Being screened as malnourished or at risk of malnutrition using the Mini Nutritional Assessment-Short Form (MNA-SF) with a score at 11 or below
* Willing to follow the study procedures
* Written informed consent form

Exclusion Criteria:

* Recent (i.e. past 3 months) or concurrent participation in any clinical trial or dietary intervention program
* Self-reported allergy or intolerance to the ingredients of the nutrition supplement
* Consumption of additional ONS, tube feeding or parenteral nutrition
* Use of medications (Amphetamine and its derivatives, Levothyroxine, Biguanides) that could affect study outcomes
* With cancer conditions that are currently undergoing treatment
* Poorly controlled or unstable chronic obstructive pulmonary disease
* Poorly controlled or unstable cardiovascular disease or diabetes or hypertension
* Recent unhealed bone fracture (within the past 12 months)
* Existing gastrointestinal (GI) diseases or pathological findings, which do not allow enteral feeding, e.g. intestinal atony, ileus, acute upper GI bleeding, shock, or malabsorption, e.g. inflammatory bowel disease, pancreatic disease, or previous surgical GI resection
* Severely impaired gastrointestinal function, i.e. severe constipation or acute diarrhea (≥ 3 loose or watery stools per day)
* Dysphagia or high aspiration risk
* Long-term bedridden
* Liver failure or severe renal insufficiency (i.e. significant renal impairment at eGFR of <30 ml/min, or significant liver impairment as indicated by ALT>100 or history of liver cirrhosis) in the past 3 months before enrollment
* Relevant central nervous system and/or psychiatric disorders, i.e. Stroke, Alzheimer's disease, Parkinson's disease, traumatic brain injury, depression or other mood disorders
* Planned surgery or hospitalization during study period
* With any other indication of a major medical or psychological illness, as judged by the investigators as ineligible to participate the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
body weight | 12 weeks
  Change in body weight

SECONDARY OUTCOMES:
Body Mass Index | 12 weeks
  Change in Body Mass Index. Height will be measured twice to the nearest 0.1 cm and body weight will be measured twice to the nearest 0.1 kg. BMI will be calculated as body weight in kg / (height in m)2.
Mini Nutritional Assessment-short form(MNA-SF) | 12 weeks
  Change in MNA-SF would be used to examine the nutritional status of the participants. The scale of this test would be 0 to 14. Malnutrition or at risk of malnutrition will be classified as having a score of 11 or below. Score of 12-14 would be defined as normal nutritional status.
SF-12 Health Survey | 12 weeks
  Health-related quality of life will be measured with the validated Chinese version of SF-12, which includes physical and mental domains. Physical and Mental Health Composite Scores are computed using the scores of twelve questions and range from 0 to 100. Higher score indicates better health-related quality of life in both domains.
Self-rated health | 12 weeks
  Self-rated health will be elicited by a single question, "Generally speaking, how is your health: excellent, very good, good, fair, or poor?"The scale would 1 to 5 and a lower score indicates worse self-rated health in this study.
5-item FRAIL scale | 12 weeks
  The 5-item FRAIL scale will be measured.A score of 1 is assigned to each of the five components: fatigue, resistance (i.e. inability to climb up 10 steps), ambulation (i.e. inability to walk two to three blocks), having more than five diseases, and recent weight loss of more than 5%. Frailty scores range from 0 to 5 and represent frail (3 to 5), pre-frail (1 to 2), and robust (0) health status.
3-day dietary record | 12 weeks
  3-day dietary record will be used to capture dietary intake for 3 days. The days of recording will be randomly assigned so that all days of the week, including weekend days, will be equally represented. Instructions about recording type of foods and how to estimate the portion sizes in household measures will be given. On the scheduled visit, the trained personnel will check the dietary records for completeness, obtain additional information about unclear items or amounts, and use examples of household measures to improve the estimation. The daily nutrient intake will be calculated by the Food Processor Nutrition analysis and Fitness software version 8.0 (ESHA Research, Salem, USA), with addition of composition of local foods based on food composition table from China and Hong Kong. Change in diet quality in terms of energy intake would be measured as outcome.
mid-arm circumference (MAC) | 12 weeks
  change of MAC in cm
calf circumference | 12 weeks
  change of calf circumference in cm

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kwok, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No